CLINICAL TRIAL: NCT03432260
Title: An Open- Label, Dose Escalation Study to Assess the Safety, Pharmacokinetics and Pharmacodynamic Signals of DUR-928 in Patients With Alcoholic Hepatitis
Brief Title: A Research Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of DUR-928 in Patients With Alcoholic Hepatitis
Acronym: AH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C928-010
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2022-11

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; acute alcoholic liver disease; progressive inflammatory liver injury; IV infusion
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Intervention Model Description: Staggered parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Moderate AH) DUR-928 30 mg (Experimental): Lowest dose of 3 dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 30 mg
- Part A (Moderate AH) DUR-928 90 mg (Experimental): Middle dose of 3 dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 90 mg
- Part A (Moderate AH) DUR-928 150 mg (Experimental): Highest dose of dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 150 mg
- Part B (Severe AH) DUR-928 30 mg (Experimental): Lowest dose of dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 30 mg
- Part B (Severe AH) DUR-928 90 mg (Experimental): Middle dose of dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 90 mg
- Part B (Severe AH) DUR-928 150 mg (Experimental): Highest dose of dose escalation arms: 30mg, 90 mg and 150 mg
  Interventions: Drug: DUR-928 150 mg

INTERVENTIONS:
Drug: DUR-928 30 mg — Lowest dose of 3 dose escalation arms.
  Arms: Part A (Moderate AH) DUR-928 30 mg; Part B (Severe AH) DUR-928 30 mg
Drug: DUR-928 90 mg — Middle dose of 3 dose escalation arms.
  Arms: Part A (Moderate AH) DUR-928 90 mg; Part B (Severe AH) DUR-928 90 mg
Drug: DUR-928 150 mg — Highest dose of 3 dose escalation arms.
  Arms: Part A (Moderate AH) DUR-928 150 mg; Part B (Severe AH) DUR-928 150 mg

SUMMARY:
This is a research trial testing DUR-928 (an experimental medication). The purpose of this trial is to assess the dose related safety, Pharmacokinetics, and Pharmacodynamics of DUR 928 in patients with moderate and severe alcoholic hepatitis (AH).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (either from patient or patient's legally acceptable representative)
2. Male or female patients 21 years of age or older with BMI ≥ 20 to ≤ 40 kg/m2
3. Patients with alcoholic hepatitis defined as:

   1. History of heavy alcohol abuse: > 40 g/day in females or > 60 g/day in males for a minimum period of 6 months, AND
   2. Consumed alcohol within 12 weeks of entry into the study, AND
   3. Serum bilirubin > 3 mg/dL AND AST > ALT, but less than 300 U/L AND
   4. MELD score between 11-30, inclusive
4. No evidence of active infection as determined by the investigator.
5. Women of child-bearing potential must utilize appropriate birth control throughout the study duration.
6. Male patients must agree to use a medically acceptable method of contraception/birth control throughout the study duration

Exclusion Criteria:

1. Other or concomitant cause(s) of liver disease as a result of:

   1. Autoimmune liver disease
   2. Wilson disease
   3. Vascular liver disease
   4. Drug induced liver disease
2. Co-infection with human immunodeficiency virus (HIV) or Hepatitis B
3. Any active malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)
4. If female, known pregnancy, or has a positive serum pregnancy test, or lactating/breastfeeding
5. Serum creatinine > 2.5 mg/dL
6. Patients who have had organ transplantation (such as liver, kidney, lung, heart, bone marrow, or stem cell etc.), other than cornea transplant
7. Stage 3 or greater encephalopathy by West Haven criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gordon, MD, Study Director — CTI Clinical Trial and Consulting Services
Locations (7):
- United States (7):
  - DURECT Study Site 0001, San Diego, California
  - DURECT Study Site 007, Miami, Florida
  - DURECT Study Site 0004, Atlanta, Georgia
  - DURECT Study Site 0002, Chicago, Illinois
  - DURECT Study Site 008, Indianapolis, Indiana
  - DURECT Study Site 0005, Louisville, Kentucky
  - DURECT Study Site 006, San Antonio, Texas

REFERENCES:
- [Derived] Hassanein T, McClain CJ, Vatsalya V, Stein LL, Flamm SL, Martin P, Cave MC, Mitchell M Jr, Barton B, Nagy L, Szabo G, McCullough A, Dasarathy S, Shah J, Blevins C, Scott D, Krebs W, Brown JE, Lin W. Safety, Pharmacokinetics, and Efficacy Signals of Larsucosterol (DUR-928) in Alcohol-Associated Hepatitis. Am J Gastroenterol. 2024 Jan 1;119(1):107-115. doi: 10.14309/ajg.0000000000002275. Epub 2023 Apr 3. PMID 37011138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A (Moderate AH) and Part B (Severe AH) were assigned treatments in a dose escalation, staggered parallel design.
  Part A (Moderate AH) highest dose of dose escalation arms (150 mg) was not enrolled.
Groups:
- Moderate AH DUR-928 30 mg: Part A (Moderate AH) Lowest dose of doses investigated: 30 mg, 90 mg, 150 mg DUR-928: Dose escalation including 2 doses: 30mg and 90 mg (150 mg did not enroll)
- Moderate AH DUR-928 90 mg: Part A (Moderate AH) Middle dose of doses investigated: 30 mg, 90 mg, 150 mg DUR-928: Dose escalation including 2 doses: 30mg and 90 mg (150 mg did not enroll)
- Severe AH DUR-928 30 mg: Part B (Severe AH) Lowest dose of doses investigated: 30mg, 90 mg and 150 mg
  DUR-928: Dose escalation including 3 doses: 30mg, 90 mg and 150 mg
- Severe AH DUR-928 90 mg: Part B (Severe AH) Middle dose of doses investigated: 30mg, 90 mg and 150 mg
  DUR-928: Dose escalation including 3 doses: 30mg, 90 mg and 150 mg
- Severe AH DUR-928 150 mg: Part B (Severe AH) Highest dose of doses investigated: 30mg, 90 mg and 150 mg
  DUR-928: Dose escalation including 3 doses: 30mg, 90 mg and 150 mg
Period: Overall Study
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Started | 4 | 3 | 4 | 4 | 4
Completed | 3 | 2 | 4 | 4 | 3
Not Completed | 1 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.5 [33.0 to 39.5] | 42.0 [33.0 to 43.0] | 45.0 [37.5 to 52.5] | 43.5 [40.0 to 45.0] | 40.5 [35.5 to 46.0] | 41.0 [35.0 to 45.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 2 | 8
  Male | 1 | 2 | 3 | 3 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 2 | 2 | 7
  Not Hispanic or Latino | 3 | 3 | 2 | 2 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 4 | 4 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 4 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Lille Model for Alcoholic Hepatitis Score
Description: The Lille score predicts response of AH subjects to treatment with glucocorticoids, such as prednisolone. This score is based on age, serum albumin, creatinine, PT, and the difference in bilirubin between pre-treatment and Day 7 post-treatment. The Lille score ranges from 0.01 to 1.00. A score >0.45 predicts a higher risk of death and the recommendation to stop steroid administration.
  Lille Score = Exp(-R)/(1 + Exp(-R))
  Where:
  R = [3.19 - (0.101 x Age in years)] + (1.47 x Albumin in g/dL) + [0.28215 x (Bilirubin initial - Bilirubin day 7 in mg/dL)] - (0.206 x Creatinine in mg/dL) - (0.11115 x Bilirubin initial in mg/dL) - (0.0096 x PT in seconds) NOTE: When calculating Lille, use "baseline" values for ALL parameters EXCEPT bilirubin at Day 7. Baseline would be the Day 1 Pre-dose sample result, if available. If not available, then use the Screening sample result.
Time Frame: Day 7
Population: ITT
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
score on a scale | 0.020 [0.01 to 0.04] | 0.050 [0.01 to 0.05] | 0.155 [0.05 to 0.19] | 0.195 [0.04 to 0.24] | 0.420 [0.08 to 0.87]

2. Primary Outcome: Model for End Stage Liver Disease (MELD) Score
Description: The MELD score at enrollment is a good predictor for AH patient prognosis. Laboratory values for international normalized ratio (INR), serum creatinine (sCr) and bilirubin are used to calculate the MELD score. The MELD score ranges from 6.0 to 40.0 (capped) with a higher score predicting a higher risk of death. A sequentially improving MELD score is associated with a better chance of recovery.
  MELD score will be calculated using the original formula (pre-2016) which does not include serum sodium level.
  Original MELD Score = (0.957 x Ln(Serum Creatinine in mg/dL) + 0. 378 x Ln(Serum Bilirubin in mg/dL) + 1.120 x Ln (INR) + 0.643) x 10 Note: (1) If patient received two or more dialysis treatments within the prior 7 days, then the value for serum creatinine will be set to 4.0. (2) If any laboratory value is less than 1.0, the value will be set to 1.0 for the MELD score calculation, in order to avoid negative values resulting from taking the natural log of values less than 1.
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7 and Day 28
Population: ITT, baseline was defined as the last non-missing value prior to study drug administration, at Screening or Day 1 Pre-dose
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
score on a scale
  Screening | 19.5 [15 to 20] | 19.0 [14 to 21] | 24.5 [21 to 28] | 24.5 [21 to 28] | 25.0 [23 to 27]
  Day 1 Pre-dose: number analyzed (Participants) | 0 | 1 | 3 | 1 | 3
  Day 1 Pre-dose |  | 20.0 [20 to 20] | 23.0 [21 to 26] | 24.0 [24 to 24] | 23.0 [21 to 26]
  Day 7: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
  Day 7 | 17.0 [16 to 19] | 17.0 [11 to 19] | 23.5 [21 to 29] | 24.0 [21 to 29] | 24.0 [21 to 28]
  Day 28: number analyzed (Participants) | 3 | 2 | 4 | 4 | 3
  Day 28 | 15.0 [12 to 20] | 11.5 [8 to 15] | 19.0 [16 to 24] | 23.5 [17 to 28] | 23.0 [19 to 29]

3. Primary Outcome: Model for End Stage Liver Disease (MELD) Score - Percent Change From Baseline
Description: The MELD Score %change from baseline is a %change between 2 time points, baseline and value at a specific time point (Day 7 or Day 28). MELD score is a good predictor of outcome. A declining MELD score suggests disease improvement. Lab values for international normalized ratio (INR), serum creatinine (sCr) and bilirubin are used to calculate the MELD score. MELD score will be calculated using the original formula (pre-2016) which does not include serum sodium level. Original MELD Score = (0.957 x Ln(Serum Creatinine in mg/dL) + 0. 378 x Ln(Serum Bilirubin in mg/dL) + 1.120 x Ln (INR) + 0.643) x 10 Note: (1) If patient received two or more dialysis treatments within the prior 7 days, then the value for serum creatinine will be set to 4.0. (2) If any laboratory value is less than 1.0, the value will be set to 1.0 for the MELD score calculation, in order to avoid negative values resulting from taking the natural log of values less than 1.
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7 and Day 28
Population: ITT
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
Percent Change
  Day 7 | -5.00 [-10.5 to 6.7] | -10.53 [-21.4 to -5.0] | 0.00 [-8.7 to 3.6] | 0.00 [-4.0 to 3.6] | 0.00 [-4.3 to 3.7]
  Day 28: number analyzed (Participants) | 3 | 2 | 4 | 4 | 3
  Day 28 | -20.00 [-21.1 to 0.00] | -33.93 [-42.9 to -25.0] | -26.76 [-35.7 to 14.3] | -8.00 [-19.0 to 8.3] | 0.00 [-29.6 to 11.5]

4. Secondary Outcome: Serum Cytokeratin 18 (M30)
Description: Analysis Population Description: Baseline was defined as the last non-missing value prior to study drug administration, at Screening or Day 1 Pre-dose.
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7, Day 28
Population: Number analyzed is dependent on samples being collected and evaluable.
Measure: Median (Full Range); unit: U/L
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
U/L
  Day 1-Predose: number analyzed (Participants) | 4 | 3 | 4 | 4 | 3
  Day 1-Predose | 723.5 [334 to 2255] | 737 [467 to 4000] | 1443.5 [561 to 4000] | 1946 [292 to 4000] | 931 [752 to 1766]
  Day 7: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
  Day 7 | 526 [257 to 3150] | 3112 [2124 to 3440] | 3305.5 [500 to 4000] | 1702.0 [323 to 4000] | 1012.5 [439 to 4000]
  Day 28: number analyzed (Participants) | 0 | 2 | 4 | 4 | 3
  Day 28 |  | 2205.5 [411 to 4000] | 1114.0 [612 to 3160] | 550.5 [243 to 4000] | 161.0 [108 to 4000]

5. Secondary Outcome: Serum Cytokeratin 18 (M65)
Description: as for outcome 4
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7, Day 28
Population: Number analyzed is dependent on samples being collected and evaluable.
Measure: Median (Full Range); unit: U/L
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
U/L
  Day 1-Predose: number analyzed (Participants) | 4 | 3 | 4 | 4 | 3
  Day 1-Predose | 252.5 [217 to 2074] | 1791.0 [729 to 14208] | 3033.5 [750 to 20000] | 4071.5 [225 to 20000] | 1999.0 [1777 to 2209]
  Day 7: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
  Day 7 | 353.0 [119 to 3029] | 4697.0 [4416 to 9928] | 7303.0 [709 to 20000] | 4397.5 [234 to 20000] | 3994.5 [502 to 15028]
  Day 28: number analyzed (Participants) | 0 | 2 | 4 | 4 | 3
  Day 28 |  | 4771.5 [807 to 8736] | 2426.0 [998 to 7420] | 1224.5 [224 to 17232] | 1987.0 [452 to 3246]

6. Secondary Outcome: International Normalized Ratio (INR) - Percent Change From Baseline
Description: ITT population. INR (international normalized ratio) is a standardized number based on the prothrombin time and calculated by the clinical lab. INR measures the time it takes for blood to clot in vitro and measures, among other things, liver synthetic function.
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7, Day 28
Population: Baseline is defined as the last non-missing value prior to study drug administration, at Screening or Day 1 Pre-dose
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
Percent Change
  Day 7 Percent Change from Baseline: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
  Day 7 Percent Change from Baseline | -10.000 [-11.11 to 7.35] | -3.226 [-8.33 to 7.14] | 4.768 [-8.88 to 10.53] | 0.000 [-5.26 to 43.75] | 0.000 [-8.33 to 6.67]
  Day 28 Percent Change from Baseline: number analyzed (Participants) | 3 | 2 | 4 | 4 | 3
  Day 28 Percent Change from Baseline | -3.676 [-22.22 to 0.00] | 0.000 [0.00 to 0.00] | -19.402 [-29.68 to 17.65] | -3.180 [-21.05 to 18.75] | 0.000 [-33.33 to 42.11]

7. Secondary Outcome: Bilirubin - Percent Change From Baseline
Description: ITT population
Time Frame: Baseline (Screening or Day 1 Pre-dose), Day 7, Day 28
Population: Baseline is defined as the last non-missing value prior to study drug administration, at Screening or Day 1 Pre-dose
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
Percent Change
  Day 7 Percent Change from Baseline: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4
  Day 7 Percent Change from Baseline | -15.69 [-34.5 to 17.1] | -31.03 [-43.9 to -29.3] | -25.19 [-49.8 to -9.0] | -6.48 [-25.1 to 6.6] | 4.96 [-29.3 to 24.7]
  Day 28 Percent Change from Baseline: number analyzed (Participants) | 3 | 2 | 4 | 4 | 3
  Day 28 Percent Change from Baseline | -27.27 [-40.0 to -5.9] | -74.27 [-75.6 to -72.9] | -56.93 [-74.1 to 34.0] | -34.82 [-47.9 to 50.0] | -10.04 [-63.6 to 1.5]

8. Other Pre Specified Outcome: Serum Creatinine (sCR)
Description: Serum Creatinine (sCR) at baseline is provided as part of the calculation for MELD
Time Frame: Baseline (Screening or Day 1 Pre-dose)
Population: Baseline was defined as the last non-missing value prior to study drug administration, at Screening or Day 1 Pre-dose.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
mg/dL
  Baseline (Screening) | 0.620 [0.46 to 0.80] | 0.710 [0.2 to 0.84] | 0.795 [0.63 to 1.20] | 0.765 [0.59 to 1.50] | 0.610 [0.50 to 1.00]
  Baseline (Day 1-Pre dose): number analyzed (Participants) | 0 | 1 | 3 | 1 | 3
  Baseline (Day 1-Pre dose) |  | 0.660 [0.66 to 0.66] | 0.640 [0.61 to 0.78] | 0.580 [0.58 to 0.58] | 0.520 [0.50 to 0.70]

ADVERSE EVENTS:
Time Frame: 28 days
Description: If subject was not available in person, they were contacted via phone.
Arm/Group | Moderate AH DUR-928 30 mg | Moderate AH DUR-928 90 mg | Severe AH DUR-928 30 mg | Severe AH DUR-928 90 mg | Severe AH DUR-928 150 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 2/4 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 3/4 | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate AH DUR-928 30 mg (N=4) | Moderate AH DUR-928 90 mg (N=3) | Severe AH DUR-928 30 mg (N=4) | Severe AH DUR-928 90 mg (N=4) | Severe AH DUR-928 150 mg (N=4)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate AH DUR-928 30 mg (N=4) | Moderate AH DUR-928 90 mg (N=3) | Severe AH DUR-928 30 mg (N=4) | Severe AH DUR-928 90 mg (N=4) | Severe AH DUR-928 150 mg (N=4)
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a joint publication is not submitted within 18-24 months after study completion, PI shall have the right to submit to sponsor a proposed results communication based on results at their institution. Sponsor can review proposed results communications prior to public release, can request removal of confidential information, and can embargo communications regarding trial results for up to 120-180 days after submission to sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03432260/Prot_SAP_001.pdf